CLINICAL TRIAL: NCT03757507
Title: Investigation of Plaque Instability: Identification of Atherosclerotic Plaque Angiogenesis Using Bevacizumab-800CW and Optoacoustic Imaging: a Single Center Proof of Concept Study (CAROTID-OPTOLIGHT)
Brief Title: Investigation of Plaque Instability Using Bevacizumab-800CW and MSOT
Acronym: Carotid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: G.M. van Dam (Other)
Responsible Party: Sponsor-Investigator, G.M. van Dam, Professor van Dam, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 201800515
Record Dates: First submitted 2018-11-26; First posted 2018-11-29 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Atherosclerosis; Carotid Stenosis; Fluorescence
MeSH Terms: conditions — Atherosclerosis; Carotid Stenosis

STUDY DESIGN:
Intervention Model Description: Open label, single group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optoacoustic imaging (Experimental): Optoacoustic Imaging before and after tracer administration
  Interventions: Device: MultiSpectral Optoacoustic Tomography

INTERVENTIONS:
Device: MultiSpectral Optoacoustic Tomography — Multispectral Optoacoustic Tomography is a new emerging imaging technique which uses laser light to heat up molecules with a high pulsed laser. The molecules undergo thermal expansion and produces sound waves, which can be detected by special transducers. The device can pick up different signals in different wavelength to produce images with anatomic and biological information.

SUMMARY:
Determining whether we could visualize uptake of the fluorescent tracer Bevacizumab-800CW, targeting VEGF-A in atherosclerotic plaques by using the new imaging technique Multispectral Optoacoustic Tomography both in- and ex vivo.

DETAILED DESCRIPTION:
Rationale: This project consists of the realization followed by the clinical validation of a procedure dedicated to detect vulnerable atherosclerotic plaques patients with a symptomatic carotid stenosis. If in the future it would be possible to detect a symptomatic carotid atherosclerotic plaque non- invasively (i.e. those plaques resulting in cerebrovascular accidents and/or transient ischemic attacks), this would strongly improve risk assessment among this large cohort of patients. At the moment, indications for intervention are primarily based on degree of stenosis, and not on degree of vulnerability. Symptomatology is considered, but clinicians are not capable of predicting the consequences of a first event, while two thirds of all patients with a major stroke are not preceded by previous minor symptoms. Previous trials (NASCET and ECST) showed a significant absolute risk reduction for symptomatic patients with a stenotic lesion of the internal carotid artery greater than 70% after the performance of a carotid endarterectomy (CEA; excision of the atherosclerotic plaque). However, surgery can be associated with significant morbidity and even mortality. On the other hand, reliable prediction prior to surgery whether an atherosclerotic plaque is going to become symptomatic could also prevent unnecessary surgery, which again significantly reduces morbidity and mortality.

In literature and our preliminary ex vivo data with a nuclear imaging tracer 89Zr-Bevacizumab, it appears that vulnerable atherosclerotic plaques (i.e. those likely to become symptomatic) have an increased rate of angiogenesis at the site of the rupture (i.e. the site of the vulnerable plaque) which expose highly upregulated Vascular Endothelial Growth Factor-A (VEGF-A) production as part of the inflammatory response within the plaque and subsequently which can be visualized with a tracer targeting specifically VEGF-A. Recently, these experiments have been repeated using Bevacizumab- CW800 showing similar results (Huisman et al, preliminary data).

An intraoperative near-infrared fluorescence (NIRF) imaging camera, among a NIR fluorescence endoscopy system, and the use of the optical contrast agent Bevacizumab-800CW in now more than 250 patients has been evaluated for its feasibility to detect tumor lesions in patients with colorectal cancer, colon polyps, Barret's esophagus, peritoneal carcinomatosis of colorectal cancer origin and breast cancer. These studies showed that bevacizumab-800CW is safe in clinical use and feasible to detect even small tumor lesions with a high sensitivity. While Bevacizumab-800CW can also detect the soluble ligand VEGF-A, as shown by ex vivo analyses of excised CEA specimen, we aim to investigate whether systemic administered Bevacizumab-800CW can be applied to patients preoperatively for the detection of vulnerable plaques by non-invasive optoacoustic imaging and subsequently ex vivo mesoscopic imaging for validation purposes. The primary objective for the proposed study is to achieve pre-operative detection of the atherosclerotic plaque for patients with a symptomatic carotid artery stenosis by non-invasive optoacoustic imaging. In this study we will introduce the following concept: a preoperative non-invasive optoacoustic-scan guided by the © UMCG october 2018 Version 2.0 7 of 40

Bevacizumab-800CW targeted VEGF-A. This will help us to detect if and at what time point within the atherosclerotic plaque there is an upregulation of angiogenesis which can cross-correlated by ex vivo analyses of characteristics of the vulnerable plaque (i.e. atheroma, foam cells, influx of activated macrophages and angiogenesis as a result of pro-inflammatory responses present in the plaque). The end-goal of the proposed dual pre- and intra-operative imaging procedure is to prove that the symptomatic carotid atherosclerotic plaque can be accurately and safely detected by VEGF-A targeted optical imaging agents. In addition, this study serves as a step-up to a larger non-invasive VEGF-A targeted optical imaging study expanding the detection technology by using a new non- invasive multispectral optoacoustic detection system. Ultimately, VEGF-A targeted imaging in carotid stenosis could be used to predict vulnerability of the atherosclerotic plaque non-invasively in order to select those patients who will benefit the most of a surgical procedure.

Objective:

This feasibility study has two objectives:

* To investigate whether it's feasible to detect plaques within the carotid artery using optoacoustic imaging with the innovative MSOT Acuity Echo in patients with symptomatic carotid stenosis.
* To investigate whether the VEGF-targeted optical imaging agent Bevacizumab-800CW is able to detect VEGF upregulation as a characteristic of the vulnerable plaque in carotid tissue by means of pre-operative Bevacizumab-800CW optoacoustic imaging in patients with symptomatic carotid stenosis cross-correlated by ex vivo histopathological analyses.

Study design: Interventional phase 1 technical feasibility study: non-randomized, open label, uncontrolled with single group proof of concept study. This study will be carried out at the University Medical Center Groningen, Department of Surgery and Department of Nuclear Medicine and Molecular Imaging. Further analysis of sections of the plaques will be done at the Department of Pathology at the UMCG and by the Helmholtz Institute, Biomedical Research Centre, München.

Study population: Patients planned for elective endarterectomy for symptomatic carotid stenosis will undergo prior to surgery imaging with an optoacoustic device before and after intravenous injection with the VEGF-targeted optical imaging agent Bevacizumab-800CW.

Intervention: Patients planned to undergo endarterectomy for symptomatic carotid stenosis will be consented for this study. The procedure will in no way delay the time interval between onset of symptoms and intervention. Three days before the planned fluorescent optoacoustic scanning, the patients will undergo optoacoustic imaging as a reference. Patients then receive an intravenous injection of 4,5 mg flat-dose of Bevacizumab-800CW. Three days after tracer administration, mostly

© UMCG october 2018 Version 2.0 8 of 40

the day patients are admitted to the hospital as standard-of-care, patients will undergo final optoacoustic imaging.

Main study parameters/endpoints:

Primary Objective:

* Feasibility of optoacoustic imaging to image the carotid artery and detect plaque formation in patients with symptomatic carotid artery disease.
* Pre-operative detection of the atherosclerotic plaque in symptomatic carotid stenosis by the VEGF-targeted optical imaging agent optical imaging agent Bevacizumab-800CW using optoacoustic imaging subsequently correlated ex vivo for VEGF upregulation within the plaque indicative for increased angiogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 21 with an indication to undergo a carotid endarterectomy for suspected symptomatic atherosclerotic plaque based on the presence of a CVA and/or transient ischemic attacks (TIA's), including amourosis fugax.

  1. Patients with significant and symptomatic carotid stenosis who are scheduled for carotid endarterectomy as decided by the surgeon or the Multi-Disciplinary Carotid Board

Exclusion Criteria:

1. Medical or psychiatric condition that compromises the patient's ability to give informed consent
2. Pregnant or lactating women
3. Significantrenal(creatinine>110μmol/L)dysfunction
4. History of iodine allergy or anaphylactic reactions to insect bites or medication or previous allergic reaction to bevacizumab
5. Presence or history of hyperthyroidism

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-04-10 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of MSOT imaging | 12 months
  Feasibility of optoacoustic imaging to image the carotid artery and detect plaque formation in patients with symptomatic carotid artery disease.
Ex vivo imaging | 12 months
  Pre-operative detection of the atherosclerotic plaque in symptomatic carotid stenosis by the VEGF-targeted optical imaging agent optical imaging agent Bevacizumab-800CW using optoacoustic imaging subsequently correlated ex vivo for VEGF upregulation within the plaque indicative for increased angiogenesis.

SECONDARY OUTCOMES:
Location of Fluorescence | 12 months
  Presence of fluorescent signaling after excision of the atherosclerotic plaque ex vivo as determined by flatbed scanning and fluorescence microscopy.

IPD SHARING:
Plan to Share IPD: Undecided